CLINICAL TRIAL: NCT02097004
Title: Phase4, to Compare Efficacy and Safety of Therapeutic Vaccination With Intensified Schedule Plus Pegylated Interferon Dual Therapy on Seroclearance of HBS Antigen in Patients With Complete Virological Response Induced by Entecavir
Brief Title: Study of Therapeutic Vaccination With Intensified Schedule Plus Pegasys Dual Therapy on Chronic Hepatitis B Infection
Acronym: E+VIP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yoon Jun Kim, MD, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E+VIP
Record Dates: First submitted 2014-03-23; First posted 2014-03-26 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis B, Chronic
Keywords: chronic hepatitis B; Pegasys; Euvax B; Baracrude
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Concomitant:Pegasys, Euvax B, Baracrude (Experimental): * Peginterferon alfa-2a: once weekly 180 μg subcutaneous injection for 48 weeks
  * HBV vaccination (Euvax B Inj): 1.0 mL (20 μg) intramuscular injection at 4, 8, 12 and 28 weeks
  * Continue Entecavir(0.5mg) for 100 weeks(once daily)
  Interventions: Biological: Peginterferon alfa-2a; Biological: HBV vaccination; Drug: Entecavir
- Sequential:Pegasys, Euvax B, Baracrude (Experimental): * Peginterferon alfa-2a: once weekly 180 μg or weight base dose subcutaneous injection for 48 weeks
  * HBV vaccination (Euvax B Inj): 1.0 mL (20 μg) intramuscular injection at 52, 56, 60 and 76 weeks
  * Continue Entecavir(0.5mg) for 100 weeks(once daily)
  Interventions: Biological: Peginterferon alfa-2a; Biological: HBV vaccination; Drug: Entecavir
- Control Group (Active Comparator): * Continue Entecavir(0.5mg) for 100 weeks(once daily)
  * After EOS(100W), injection(once weekly) a Peginterferon alfa-2a for 48 weeks
  Interventions: Biological: Peginterferon alfa-2a; Drug: Entecavir

INTERVENTIONS:
Biological: Peginterferon alfa-2a — once weekly 180 μg subcutaneous injection for 48 weeks
  Other Names: Pegasys
Biological: HBV vaccination — 1.0 mL (20 μg) intramuscular injection at 4, 8, 12 and 28 weeks
  Other Names: Euvax B Inj
  Arms: Concomitant:Pegasys, Euvax B, Baracrude; Sequential:Pegasys, Euvax B, Baracrude
Drug: Entecavir — Continue Entecavir(0.5mg) for 100 weeks
  Other Names: Baracrude

SUMMARY:
A randomized, Open label, Single center, Prospective study to compare efficacy and safety of Therapeutic Vaccination with Intensified schedule plus Pegylated Interferon dual Therapy on Seroclearance of Hepatitis B virus Surface Antigen in Patients with Complete Virological Response Induced by Entecavir

DETAILED DESCRIPTION:
A randomized, Open label, Single center, Prospective study to compare efficacy and safety of Therapeutic Vaccination with Intensified schedule plus Pegylated Interferon dual Therapy on Seroclearance of Hepatitis B virus Surface Antigen in Patients with Complete Virological Response Induced by Entecavir (E + VIP)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 75 year-old
2. HBsAg-positive for > 6 months apart (medical history can be alternative)
3. Currently being treated with entecavir 0.5 mg/day for more than 18 months
4. Undetectable HBV DNA in serum (<20IU/mL) and HBeAg-negative or positive for > 1year
5. HBsAg titer < 3,000 IU/mL
6. ALT<300 IU/L
7. Signed written informed consent after being instructed about the objective and procedure of the clinical study

Exclusion Criteria:

1. Patients with decompensated liver cirrhosis, any one of the following ① Serum bilirubin > 3 mg/dL

   ② Prothrombin time > 6 seconds prolonged or INR >2.3

   ③ Serum albumin < 2.8 g/dL

   ④ History of ascites, variceal hemorrhage, or hepatic encephalopathy

   ⑤ Child-Pugh score ≥7 (Child-Pugh class B or C)
2. Patients who have evidence of renal insufficiency defined as serum creatinine>1.5 mg/dL
3. Patients with psychological problem including depression
4. Patients who have previous/current significant co-morbidities including congestive heart failure, chronic kidney disease, hematologic disease and malignancy including hepatocellular carcinoma(patients with malignancy cured 5 years before screening can be enrolled)
5. Patients with seropositivity for anti-HCV, anti-HDV or anti-HIV
6. Patients who have excessive alcohol consumption (> 30 g/day)
7. Patients who have evidence of autoimmune hepatitis, hemochromatosis or Wilson's disease
8. Pregnant or breast feeding females or plan for pregnancy or no contraception
9. Patients with disease may deteriorate with interferon therapy(eg, autoimmune thyroiditis)
10. Patients who have an psoriasis
11. Patients who have history of antiviral-resistant HBV after previous treatment with oral antiviral agents
12. Previous diagnosis with immunodeficiency or concomitant treatment of immune suppressive agent or previous organ transplantation Recipients
13. Patients who have a history of hypersensitivity to study drug
14. Uncontrollable seizure, convulsion and/or central nervous system disorders
15. Patients with severe bone marrow disorder or with history of hypersensitivity to biologic agent such as vaccine.
16. Neutrophil count < 1,500/mm3 or platelet count < 75,000/mm3 or hemoglobin < 10 g/dl
17. Patients with Pulmonary disease (in case of history of pulmonary disease with complete recovery, enrollment is on investigator's discretion)
18. Patients who have a fever ≥ 38 °C at the baseline
19. Patients who have a risk of febrile response or systemic reaction
20. Patients who the investigator deems inappropriate to participate in this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
The rate of HBsAg-seroclearance | The rate of HBsAg-seroclearance at the time point of at weeks 100
  The rate of HBsAg-seroclearance at the time point of at weeks 100 in the sequential treatment group (24 weeks after termination of treatment) versus control group(ETV monotherapy) at weeks 100.

SECONDARY OUTCOMES:
The rate of HBsAg-seroconversion | The rate of HBsAg-seroconversion at weeks 100
  The rate of HBsAg-seroconversion at weeks 100 in the sequential treatment group versus control group(ETV monotherapy) at weeks 100.
The change of HBsAg level from baseline | The change of HBsAg level from baseline at weeks 100
  The change of HBsAg level from baseline at weeks 100 in the sequential treatment group versus control group(ETV monotherapy) at weeks 100.
The change of HBsAg-seroclearance | The change of HBsAg-seroclearance at weeks 4, weeks 12, weeks 24, weeks 36, weeks 48, weeks 60, weeks 72, weeks 96, weeks 100, weeks 148
  The change of HBsAg-seroclearance in the concomitant treatment group versus control group(ETV monotherapy) for exploratory assessment.
The change of HBsAg-seroconversion | The change of HBsAg-seroconversion at weeks 4, weeks 12, weeks 24, weeks 36, weeks 48, weeks 60, weeks 72, weeks 96, weeks 100, weeks 148
  The change of HBsAg-seroconversion in the concomitant treatment group versus control group(ETV monotherapy) for exploratory assessment.
The change of HBsAg level | The change of HBsAg level at weeks 4, weeks 12, weeks 24, weeks 36, weeks 48, weeks 60, weeks 72, weeks 96, weeks 100, weeks 148
  The change of HBsAg level in the concomitant treatment group versus control group(ETV monotherapy) for exploratory assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Jun Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Lee YB, Cho EJ, Yu SJ, Yoon JH, Kim YJ. Entecavir Plus Pegylated Interferon and Sequential Hepatitis B Virus Vaccination Increases Hepatitis B Surface Antigen Seroclearance: A Randomized Controlled Proof-of-Concept Study. Clin Infect Dis. 2021 Nov 2;73(9):e3308-e3316. doi: 10.1093/cid/ciaa807. PMID 32556157